CLINICAL TRIAL: NCT02487628
Title: Multi-center, Randomized, Active-controlled, Single-blind, Parallel Two-group Trial of HQ® Matrix Soft Tissue Mesh and ULTRAPRO® Partially Absorbable Lightweight Mesh for the Treatment of Inguinal Hernia
Brief Title: Evaluation of HQ® Matrix Soft Tissue Mesh for the Treatment of Inguinal Hernia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Xingyue Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: YL-QX-YYZZBP-2014
Record Dates: First submitted 2015-06-26; First posted 2015-07-01 (Estimated); Last update posted 2015-07-01 (Estimated); Status verified 2015-06

CONDITIONS: Inguinal Hernia
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HQ® Matrix Soft Tissue Mesh (Experimental): HQ® Matrix Soft Tissue Mesh is a warp-knitted, multifilament, bioengineered scaffold which is comprised of the silk fibroin protein of the Bombyx mori (B. mori) silkworm. The porous network structure makes it soft and pliable and convenient to implant. The mesh is mechanically strong, biocompatible, and long-term bioresorbable. The pore size is suitable for macrophage migration and recruitment, which hinders bacteria growth. The mesh is provided in single sheets of varying widths and lengths and may be cut to the shape or size desired for a specific application. It is sterile and for single-patient use only.
  Interventions: Device: HQ® Matrix Soft Tissue Mesh
- ULTRAPRO® Partially Absorbable Lightweight Mesh (Active Comparator): ULTRAPRO® Partially Absorbable Lightweight Mesh (Ethicon, Inc.) is manufactured from approximately equal parts of absorbable poliglecaprone-25 monofilament fiber and non-absorbable polypropylene monofilament fiber. Designed for open and laparoscopic hernia repairs, it allows surgeons the versatility to perform various hernia repairs with a single technology. It offers excellent strength with minimal foreign body mass, to allow patients to heal more naturally with increased comfort and mobility.
  Interventions: Device: ULTRAPRO® Partially Absorbable Lightweight Mesh

INTERVENTIONS:
Device: HQ® Matrix Soft Tissue Mesh
  Other Names: HQ® Matrix
  Arms: HQ® Matrix Soft Tissue Mesh
Device: ULTRAPRO® Partially Absorbable Lightweight Mesh
  Other Names: ULTRAPRO®
  Arms: ULTRAPRO® Partially Absorbable Lightweight Mesh

SUMMARY:
The purpose of the study is to evaluate the safety and effectiveness of HQ® Matrix Soft Tissue Mesh for the Treatment of Inguinal Hernia. Half of participants will receive HQ® Matrix Soft Tissue Mesh, while the other half will receive ULTRAPRO® Partially Absorbable Lightweight Mesh.

DETAILED DESCRIPTION:
HQ® Matrix Soft Tissue Mesh is a warp-knitted, multifilament, bioengineered scaffold which is comprised of the silk fibroin protein of the Bombyx mori (B. mori) silkworm. The porous network structure makes it soft and pliable and convenient to implant. The mesh is mechanically strong, biocompatible, and long-term bioresorbable. The pore size is suitable for macrophage migration and recruitment, which hinders bacteria growth. The mesh is provided in single sheets of varying widths and lengths and may be cut to the shape or size desired for a specific application. It is sterile and for single-patient use only.

ULTRAPRO® Partially Absorbable Lightweight Mesh (Ethicon, Inc.) is manufactured from approximately equal parts of absorbable poliglecaprone-25 monofilament fiber and non-absorbable polypropylene monofilament fiber. Designed for open and laparoscopic hernia repairs, it allows surgeons the versatility to perform various hernia repairs with a single technology. It offers excellent strength with minimal foreign body mass, to allow patients to heal more naturally with increased comfort and mobility.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed clinically as inguinal hernia;
2. Need to be treated with open tension-free hernioplasty;
3. BMI ≤ 40 kg/m^2;
4. Aged from 18 - 70, male or female;
5. The patients voluntarily signed the subjects' informed consent form.

Exclusion Criteria:

1. Surgeries that cut the gastrointestinal tract or the gastrointestinal tract ruptures accidently;
2. Surgeries that repair the inguinal hernia intraperitoneally;
3. Patients that have done the hernioplasty earlier and undergone multiple recurrence (recurrence rate ≥ 2);
4. The surgical wounds are contaminated;
5. Patients that are treated with coagulant;
6. Patients with serious complication;
7. Patients with pregnancy or lactation;
8. Patients with mental disease including serious hysteria.Do not have legal capacity or have restricted capacity;
9. Those allergic to the test products;
10. Patients that participated other clinical trials in the last 3 months;
11. Patients who, according to other doctors' opinion, are unsuitable to use this material for the treatment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2014-11; Primary Completion 2016-06 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Postoperative recurrent rate | Day 1 post-operation
Postoperative recurrent rate | Day 3 post-operation
Postoperative recurrent rate | 1 day before hospital discharge
Postoperative recurrent rate | 6 months ± 14 days post-operation

SECONDARY OUTCOMES:
Number of Participants with Postoperative Complications | Day 1 and day 3 post-operation, 1 day before hospital discharge, and 6 months ± 14 days post-operation
Number of Participants with Discomfort | Day 1 and day 3 post-operation, 1 day before hospital discharge, and 6 months ± 14 days post-operation
Number of Participants with Foreign Body Sensation | Day 1 and day 3 post-operation, 1 day before hospital discharge, and 6 months ± 14 days post-operation
The average hospitalization time | 1 day before hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Jianhua Huang, Principal Investigator — Xiangya Hospital of Centre-South University
Locations (7):
- China (7):
  - Huanggang Central Hospital, Huanggang, Hubei
  - Huangshi Central Hospital, Huangshi, Hubei
  - Xiangyang Central Hospital, Xiangyang, Hubei
  - The Forth Hospital of Changsha, Changsha, Hunan
  - Xiangya Hospital of Centre-South University, Changsha, Hunan
  - Xiangtan Central Hospital, Xiangtan, Hunan
  - Taian Chinese Medicine Hospital, Taian, Shandong